CLINICAL TRIAL: NCT03914118
Title: An Examination of the Effects of Modafinil (Provigil) or Placebo on Neurocognitive Testing After General Anesthesia for Non-Cardiac Surgery in an Older Population
Brief Title: Modafinil to Prevent Postoperative Cognitive Decline
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Ronak Desai, DO, Director, Division of Regional Anesthesia, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-086
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Preoperative modafinil + postoperative placebo (Active Comparator)
  Interventions: Drug: Preoperative modafinil + postoperative placebo
- Preoperative modafinil + postoperative modafinil (Active Comparator)
  Interventions: Drug: Preoperative modafinil + postoperative modafinil
- Preoperative placebo + postoperative placebo (Placebo Comparator)
  Interventions: Drug: Preoperative placebo + postoperative placebo
- Control group (No Intervention)

INTERVENTIONS:
Drug: Preoperative modafinil + postoperative placebo — 200 mg modafinil pre-operatively and placebo immediately post-operatively.
  Arms: Preoperative modafinil + postoperative placebo
Drug: Preoperative modafinil + postoperative modafinil — 200 mg modafinil pre-operatively and 200 mg modafinil immediately post-operatively.
  Arms: Preoperative modafinil + postoperative modafinil
Drug: Preoperative placebo + postoperative placebo — Placebo pre-operatively and placebo immediately post-operatively.
  Arms: Preoperative placebo + postoperative placebo

SUMMARY:
Postoperative cognitive dysfunction is a well-recognized complication of surgery. The aim of the study is to investigate whether cognitive dysfunction is reduced by the use of modafinil as shown by neurocognitive testing.The treatment effects will be evaluated compared to placebo as well as a non-surgical group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I or II
* Elective surgery
* Surgery requiring general anesthesia

  4.) Control Group will be-females & males 65 and older not scheduled for any surgical procedures for at least a 3 month period.

Exclusion Criteria:

* Neurosurgery
* Cardiac surgery
* Narcotic or illicit drug abuse
* Chronic opioid use
* Chronic use of anxiolytics
* History of pulmonary disease
* C02 retention
* Sleep apnea
* Obesity

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2013-01-31 (Actual); Study Completion 2013-01-31 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test (RAVLT) scores | 3 months
  Rey Auditory Verbal Learning Test (RAVLT) scores will be used to assess memory and learning ability in the auditory-verbal domain. The RAVLT begins with a list of 15 words, which an examiner reads aloud at the rate of one per second. The patient's task is to repeat all the words he or she can remember, in any order. This procedure is carried out a total of five times. Then, the examiner presents a second list of 15 words, allowing the patient only one attempt at recall. Immediately following this, the patient is asked to remember as many words as possible from the first list. For each trial a maximum score of 15 can be obtained, which would reflect excellent memory. The obtained scores per individual trial will be compared between the 4 different arms.
  The RAVLT will be administered preoperatively, immediately postoperatively in the PACU (except the non-surgical control group), at 1 week and at 3 months postoperatively.

IPD SHARING:
Plan to Share IPD: No